CLINICAL TRIAL: NCT02236910
Title: An Open Label Phase II, Registry Study of Lutetium-177 (DOTA0, TYR3) Octreotate (Lu-DOTA-TATE) Treatment in Patients with Somatostatin Receptor Positive Tumours
Brief Title: An Open Label Registry Study of Lutetium-177 (DOTA0, TYR3) Octreotate (Lu-DOTA-TATE) Treatment in Patients with Somatostatin Receptor Positive Tumours
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TX-LUT-001-London; Lu-DOTA-TATE (Other: Sponsor)
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2023-10

CONDITIONS: Neuroendocrine Carcinoma
Keywords: somatostatin receptor positive tumour
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — lutetium Lu 177 dotatate; Radiopharmaceuticals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary Therapy with Lu-DOTA-TATE (Experimental): Lu-DOTA-TATE (Lutetium-177 Octreotate) will be administered by intravenous infusion to participants who have not been previously treated with Lu-DOTA-TATE
  Interventions: Other: Lu-DOTA-TATE
- Secondary Therapy with Lu-DOTA-TATE (Experimental): Patients who have received previous treatment with Lu-DOTA-TATE (Lutetium-177 Octreotate) under the special access program are eligible to be treated in this study. Patients will receive Lu-DOTA-TATE by intravenous infusion.
  Interventions: Other: Lu-DOTA-TATE

INTERVENTIONS:
Other: Lu-DOTA-TATE
  Other Names: Lutetium-177 Octreotate; radiopharmaceutical

SUMMARY:
Lu-DOTA-TATE (Lutetium-177 octreotate) is a radiopharmaceutical that has been reported as being effective in controlling symptoms and increase quality of life; induce stable disease and extend progression free survival; induce a (good) partial remission and induce a complete remission in patients with a somatostatin receptor positive tumour.

The purpose of this study is to assess the efficacy of Lu-DOTA-TATE by measuring progression free survival and overall survival. This study will also asses the safety of Lu-DOTA-TATE, and the quality of life of the patients treated with Lu-DOTA-TATE.

DETAILED DESCRIPTION:
Neuroendocrine (NET) tumours have secretory and metabolic pathways not typically found in other cancers that can be utilized for molecular imaging and therapeutic targeting. The most important is somatostatin. Somatostatin receptors are useful tools in the diagnosis and treatment of NET tumours because the somatostatin analogue octreotate can be radiolabeled with lutetium-177 for imaging and therapy.

In selected populations of patients, radioisotope therapy in expert hands has been shown to be a safe and effective palliative therapy with stable disease, progression free survival benefit, symptom control and improvements in quality of life. Lutetium-177 (DOTA0, Tyr3) octreotate has been used in a significant number of clinical studies shown to be safe and effective as a therapeutic agent in patients with NET tumours. The investigators intend to further confirm these benefits with lutetium-177 octreotate, which could form the basis for a national registry study leading to registration of this therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

Group A: Primary therapy subjects will be included in the study if they meet all of the following general criteria:

1. Male or female ≥ 14 - 90 years of age. If female of child-bearing potential and outside of the window of 10 days since the first day of the last menstrual period, a negative pregnancy test is required.
2. Presence of somatostatin receptor positive tumour(s) (either histologically or Octreoscan image proven), with at least 1 tumour site reliably evaluable by CT or MRI of at least 1.5 cm (smallest dimension) with respect to RECIST criteria (the target lesion).
3. Presence of somatostatin receptors on (at least) the target lesion demonstrated by uptake of OctreoScan® at least equal to liver uptake within 12 weeks of enrollment.
4. Life expectancy greater than 26 weeks from enrollment.
5. Serum creatinine ≤ 130 μmol/L, and a measured glomerular filtration rate (GFR) using plasma clearance of ≥50 mL/min measured within 2 weeks of enrollment.
6. Haemoglobin concentration ≥ 90 g/L; white blood cell count (WBC) ≥ 3 x 109/L; platelets ≥ 100 x 109/L measured within 2 weeks of enrollment.
7. Liver function tests (serum albumin, total bilirubin, alanine amniotransferase (ALT),aspartate aminotransferase (AST) and alkaline phosphatase) ≤ 3 X the limit of normal.
8. Eastern Cooperative Oncology Group (ECOG) Performance Scale Score ≤ 2 measured within 2 weeks of enrollment.
9. Provide written informed consent prior to enrollment.
10. Ki 67 < 20%, unless patients has been treated with chemotherapy and lesions are stable (Ki 67 < 30%)

Group B: Secondary therapy subjects will be included in the study if they meet all of the following general criteria:

1. Male or female ≥ 14 - 90 years of age. If female of child-bearing potential and outside of the window of 10 days since the first day of the last menstrual period, a negative pregnancy test is required.
2. Have received Lu-DOTA-TATE treatment at the London Health Sciences Centre under the Special Access Programed or other radionuclide therapy for neuroendocrine tumor.
3. Provide written informed consent prior to enrollment.

Exclusion Criteria:

Group A: Primary therapy subjects will be excluded from the study if they meet any of the following criteria:

1. Potential for surgery with curative intent. Local surgery for symptomatic relief permitted as long as target lesion unaffected.
2. Surgery, radiation therapy, radioisotope therapy, change in Sandostatin LAR therapy dosage, cytotoxic chemotherapy, embolization or other investigative therapy [interferons, mammalian target of rapamycin (mTOR) inhibitors] within 12 weeks of enrollment. Localized external beam irradiation permitted as long as target lesion unaffected.
3. Known brain metastases unless these metastases have been treated or stable (confirmed by CT) for ≥ 6 months prior to enrollment
4. Uncontrolled diabetes mellitus defined as fasting glucose ≥ 3 X the upper limit of normal within 12 weeks of enrollment.
5. Another significant medical, psychiatric or surgical condition uncontrolled by treatment, which may interfere with completion or conduct of the study (such as urinary incontinence, co-existing malignancies).
6. Pregnancy.
7. Breast feeding.
8. Prior radiation therapy to more than 25% of the bone marrow.

Group B: Secondary therapy subjects will be excluded from the study if they meet any of the following criteria:

1. Another significant medical, psychiatric or surgical condition uncontrolled by treatment, which may interfere with completion or conduct of the study (such as urinary incontinence, co-existing malignancies).
2. Pregnancy.
3. Breast feeding.

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Tumour response measured by RECIST criteria | 7 years (end of study)
  Target lesions will be assigned after treatment 1 base done either the Lu-177 scan, or the CT/MRI scan within 2 weeks prior to treatment 1. Tumour response will be measured using response evaluation criteria in solid tumours (RECIST).

SECONDARY OUTCOMES:
Progression Free Survival | 7 years (end of study)
  Progression free survival will be measured from the date of enrollment to the date the target lesion progresses as per RECIST criteria, or death sue to any cause.
Quality of Life Response Changes | 7 years (end of study)
  Quality of life changes due to treatment with Lu-DOTA-TATE, measured using the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire(QLQ) EORTC QLQ-C30.

CONTACTS AND LOCATIONS:
Overall Officials: david laidley, MD, Principal Investigator — London Health Sciences Centre & Lawson Health Research Institute
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Swiha MM, Sutherland DEK, Sistani G, Khatami A, Abazid RM, Mujoomdar A, Wiseman DP, Romsa JG, Reid RH, Laidley DT. Survival predictors of 177Lu-Dotatate peptide receptor radionuclide therapy (PRRT) in patients with progressive well-differentiated neuroendocrine tumors (NETS). J Cancer Res Clin Oncol. 2022 Jan;148(1):225-236. doi: 10.1007/s00432-021-03672-w. Epub 2021 Jun 10. PMID 34110489